CLINICAL TRIAL: NCT05653206
Title: IN-TWIN: Traumatic Incomplete Tetraplegia Without Instability: a Prospective Multicenter Feasibility Study of Outcomes and Prognosis
Brief Title: Incomplete Cervical SCI Without Instability
Status: Recruiting | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: IN-TWIN
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cervical Spinal Cord Injury
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Nonsurgical treatment — Cervical collar, Halo ring, Halo vest, cervical braces, skeletal skull traction, MAP, steroids, observation or bedrest
Procedure: Surgical treatment — Anterior discectomy and instrumented fusion (single level), Anterior discectomy and instrumented fusion (multi-level), Posterior decompression-laminectomy, Posterior decompression-laminoplasty, Posterior decompression and instrumented fusion, Combined anterior and posterior decompression and instrumented fusion

SUMMARY:
A multicenter, international, prospective, observational case series patient cohort with incomplete cervical SCI without instability will be enrolled to obtain information and data that could inform the feasibility of administering a set of additional core and optional outcome assessments in cervical SCI patients to capture the aspects of neurologic impairment. Baseline, intraoperative, and postoperative characteristics, including demographics, injury details, treatment details, neurological assessments, gait and balance assessments and upper extremity assessments, will be recorded for adult patients.

DETAILED DESCRIPTION:
This prospective multicenter study will enroll 50 adult patients with acute traumatic cervical SCI with ISNCSCI AIS Grade D or sensory deficits only without biomechanical instability.

Patients will be assessed at the baseline visit and subsequently be followed up at 3 and 6 months. All decisions regarding the treatment and clinical management will be left to the attending spinal surgeon and will follow the local standard of care.

The core outcome assessments include:

* Neurological status by the ISNCSCI
* Patient-reported outcome measures (PROMs) of Short Form-36 (SF-36) v2 and Neuropathic Pain Scale (NPS)
* The Spinal Cord Independence Measure (SCIM) v3
* Gait and balance evaluated using the ten-meter walk test (10mWT) and Walking Index for Spinal Cord Injury (WISCI) v2
* Upper extremity impairment evaluated using the grip strength with digital dynamometry, pinch strength (key pinch and tip-to-tip pinch), and the Partial Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP) v2.

All core outcome assessments will be performed at the baseline, 3-, and 6-month visits except for the PROMs, SCIM v3, key pinch and tip-to-tip pinch, which will be assessed only at the 3- and 6-month visits.

The optional outcome assessment is the multiparametric quantitative spinal cord magnetic resonance imaging (MRI)/diffusion tensor imaging (DTI) which will be performed at baseline, 3-, and 6-month visits if it is done at the surgeon's discretion.

The goal of this study is to obtain information and data that could inform the feasibility of administering a set of additional core and optional outcome assessments in cervical SCI patients with incomplete tetraplegia without spinal instability to capture the aspects of neurologic impairment that may not be well represented in the ISNCSCI examination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, inclusive
* Diagnosis of acute traumatic cervical SCI with ISNCSCI AIS Grade D or sensory deficits only within 92 hours post injury
* Cervical neurological level of injury (C2-C8)
* MRI, using any imaging protocols (conventional, multiparametric, or quantitative), taken according to standard of care
* Presence of spinal cord compression on the MRI
* Absence of biomechanical instability to the extent that would mandate stabilization surgery by the treating surgeon
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Nontraumatic SCI
* Concomitant traumatic brain injury or polytrauma that could preclude accurate or reliable assessments of the outcome assessments
* Uncontrolled severe systemic diseases, preexisting neurological, musculoskeletal, or general medical conditions which could preclude accurate assessments or FUs
* Individuals unable to undergo MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic incomplete cervical SCI without instability
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of the core outcome assessments successfully completed at each visit | up to 6 months
  For baseline and each FU visit, the completion status of each core outcome assessment
Time required to complete the individual core outcome assessments | up to 6 months
  For baseline and each FU visit, the time required for completion for each core outcome assessment will be recorded (start time, end time, and duration in mins)
Total time required to complete all core outcome assessments at each visit | up to 6 months
  The time required for completion will be measured to the nearest 0.1 second by using a digital timer, and the timing should start at the start of giving instructions to the patients or explaining the tests to the patients (start time) and end when the final score of the test is obtained (end time).
Completion rate of individual core outcome assessments (and their scorings if applicable) | up to 6 months
  Completion rate of individual core outcome assessments at each visit.
Completion rate of the multiparametric quantitative spinal cord MRI/DTI | up to 6 months
  Completion rate of the multiparametric quantitative spinal cord MRI/DTI
FU visit compliance rate and reasons for non-compliance | up to 6 months
  Completion status of FU visits, recorded at 3- and 6-month visits
Patient accrual rate | up to 6 months
  Whether the patient drops out from the study, recorded at the time of dropout

SECONDARY OUTCOMES:
Results from the core outcome assessment ISNCSCI | up to 6 months
  Motor and sensory scores (motor score 0-100, pin prick score 0-112), AIS Grades, Clinical syndrome (Central Cord/Brown-Sequard/Anterior Cord/Conus Medullaris/Cauda Equina/No clinical syndrome/Not assessed)
Results from the core outcome assessment SF-36 v2 | up to 6 months
  Eight scale scores (0-100): physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, general mental health, social functioning, energy/fatigue or vitality, and general health perceptions
Results from the core outcome assessment Neuropathic pain score | up to 6 months
  Score 0-100
Results from the core outcome assessment SCIMv3 | up to 6 months
  Three subscales: Self-care (0-20), Respiration and Sphincter Management (0-40), Mobility (room and toilet, 0-40)
Results from the core outcome assessment WISCI v2 | up to 6 months
  Level of walking (score 0-20)
Results from the core outcome assessment Key pinch and tip-to-tip pinch | up to 6 months
  Pinch strength in kg
Results from the core outcome assessment GRASSP v2 | up to 6 months
  Eight subtest scores Strength (0-50), Palmar sensation (0-12), Prehension Ability (0-12), Prehension Performance (0-20)

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson Wilson, Principal Investigator — Unity Health Toronto
Locations (10):
- United States (3):
  - San Francisco General Hospital, San Francisco, California
  - UMD STC Neurosurgery Clinic, Baltimore, Maryland
  - Medical college of Winsconsine, Neurosurgery, Milwaukee, Wisconsin
- Instituto de Ortopedia E Traumatologia Do Hospital Das Clinicas Da Universidade de Sao Paulo, São Paulo, Brazil
- Canada (3):
  - St. Michael's Hospital, Toronto
  - Toronto Western Hospital University Health Network, Toronto
  - Vancouver Spine Research Program, Blusson Spinal Cord Centre, Vancouver
- BG Klinikum Murnau gGmb, BGU Murnau, Trauma Center Murnau, Murnau am Staffelsee, Germany
- Indian Spinal Injuries Centre, New Delhi, India
- Orthopaedics, Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No